CLINICAL TRIAL: NCT05896800
Title: Efficacy and Safety of Inhaled Nitric Oxide in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease: a Prospective, Single-center Clinical Trial
Brief Title: A Clinical Study of Inhaled Nitric Oxide in Moderate-to-Severe Chronic Obstructive Pulmonary Disease
Acronym: NOVEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Novlead Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-COPD-002
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Air

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low concentration group (Experimental): inhaled nitric oxide (iNO) 10ppm，≥2 hours/day for 7 days
  Interventions: Other: Inhaled nitric oxide (NO)
- High concentration group (Experimental): iNO 40ppm，≥2 hours/day for 7 days
  Interventions: Other: Inhaled nitric oxide (NO)
- Placebo group (Placebo Comparator): patient inhaled placebo treatment
  Interventions: Other: air

INTERVENTIONS:
Other: Inhaled nitric oxide (NO) — The Nitric Oxide Generation and Delivery System is used to deliver nitric oxide for inhalation therapy into the inspiratory limb of the patient breathing circuit in a way that provides a constant concentration of nitric oxide (NO), as set by the user, to the patient throughout the inspired breath.
  Arms: High concentration group; Low concentration group
Other: air — use air（21%O2）as the placebo of inhaled treatment
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the influence of exercise capacity and safety of iNO at doses of 10 ppm or 40 ppm for 2 hours per day after continuous treatment for one week, which is of great significance for finding safe and effective methods for treating COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years, ≤ 75 years;
2. Previous smoking history ≥ 10 pack-years, and had stopped smoking for one month before study entry;
3. Met the diagnosis criteria of moderate and severe COPD: a post-bronchodilator FEV1/FVC < 0.7, and 30%< FEV1 < 80% predicted;
4. Signed informed consent and performed all the study mandated procedures.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Current or recent month user of nicotine-like substances (including nicotine patches, etc.);
3. A diagnosis of asthma or other non-COPD respiratory disease, in the opinion of the Investigator;
4. Lack of patency of nares upon physical examination;
5. Experienced during the last month an exacerbation requiring start of or increase in systemic oral corticosteroid therapy;
6. Left ventricular systolic dysfunction: left ventricular ejection fraction (LVEF) < 50%;
7. Clinically significant valvular heart disease, including aortic valvular disease (moderate or severe aortic stenosis or regurgitation) and/or mitral valve disease (moderate or severe mitral stenosis or regurgitation), or status post mitral valve replacement;
8. Use within 30 days of screening or current use of approved pulmonary hypertension medications such as sildenafil, bosentan or prostacyclines;
9. Use of investigational drugs or devices within 30 days prior to enrollment into the study;
10. Any underlying medical or psychiatric condition that, in the opinion of the Investigator, makes the subject an unsuitable candidate for the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Test: Maximal oxygen uptake（VO2max） | Baseline, Day 7
  Change in VO2max from Baseline after treatment with iNO
Cardiopulmonary Exercise Test: Minute ventilation-to-carbon dioxide output（VE/VCO2） | Baseline, Day 7
  Change in VE/VCO2 from Baseline after treatment with iNO
Cardiopulmonary Exercise Test: Borg score | Baseline, Day 7
  Change in Borg score from Baseline after treatment with iNO
Cardiopulmonary Exercise Test: oxygen uptake/work (△VO2/△W) ratio | Baseline, Day 7
  Change in △VO2/△W ratio from Baseline after treatment with iNO

SECONDARY OUTCOMES:
Pulmonary function:Forced expiratory volume in 1 second（FEV1） | Baseline, Day 7
  Change in FEV1 from Baseline after treatment with iNO
Pulmonary function: Forced vital capacity （FVC） | Baseline, Day 7
  Change in FVC from Baseline after treatment with iNO
Pulmonary function：FEV1/FVC | Baseline, Day 7
  Change in FEV1/FVC from Baseline after treatment with iNO
Life quality and symptom severity questionnaires: COPD assessment test (CAT) | Baseline, Day 7
  Change in CAT scores (0-40 scores, higher scores mean a worse outcome) from Baseline after treatment with iNO
Life quality and symptom severity questionnaires: Modified Medical Research Council (mMRC) Dyspnea Scale | Baseline, Day 7
  Change in (mMRC) Dyspnea Scale scores (0-4 scores, higher scores mean a worse outcome) from Baseline after treatment with iNO
Six-minute walk test | Baseline, Day 7
  Change in exercise capacity from Baseline after treatment with iNO: the distance of six-minute walk test
Adverse events | Baseline up to Day 7
  Incidence of adverse events = Number of subjects with adverse events/Total number of subjects in treatment×100%

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No